CLINICAL TRIAL: NCT01404975
Title: Reducing Delirium After Trans-Apical Aortic Valve Replacement (TAVI): A Multifaceted Approach of Perioperative Care
Brief Title: TAVI Protocol - Paravertebral Block Study
Acronym: TAVI PVB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UHN REB #: 11-0260-B
Record Dates: First submitted 2011-06-21; First posted 2011-07-28 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-01

CONDITIONS: Aortic Valve Replacement; Aortic Stenosis
Keywords: Delirium; PVB; PCA; Opioid; Aortic Valve replacement
MeSH Terms: conditions — Aortic Valve Stenosis; Delirium | interventions — Passive Cutaneous Anaphylaxis; PVB protocol; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paravertebral Block (Experimental): Patients randomized to receive PVB will have a continuous thoracic paravertebral block using local anesthetic after trans-apical aortic valve replacement. The patient will be placed in lateral decubitus position and under aseptic conditions the skin entry points will be 2.5-3cm from the spinal processes of the vertebra at a level of the proposed surgical incision. A 17G Touhy needle will be inserted perpendicular to the skin until the transverse process is contacted. After negative aspiration test an initial bolus of 8ml of plain ropivacaine 0.5% will be administered. This will be followed by a continuous infusion of 0.2% ropivacaine at 10 mL/hr. For break through pain additional doses of ropivacaine will be administered as required.
  Interventions: Other: Thoracic paravertebral block (PVB)
- Standard intravenous opioid analgesia (Active Comparator): Patient Controlled Analgesia (PCA) :
  PCA: the patients who are randomized to PCA group will receive standard of care for this modality.
  Interventions: Other: Thoracic paravertebral block (PVB)

INTERVENTIONS:
Other: Thoracic paravertebral block (PVB) — We are planning to replace the standard intravenous opioid analgesia with a continuous paravertebral block using local anesthetic after trans-apical aortic valve replacement.
  Anesthesia management will be standardized to minimize any impact that anesthetic type may have on neurological outcomes.
  Adjuvant supplemental analgesia will be provided to both groups according to the standardized institutional guidelines.
  Other Names: PCA, PVT, PVB, TAVI

SUMMARY:
Trans-apical aortic valve replacement is a new treatment for severe aortic stenosis. It is offered to elderly patients with medical problems that would markedly increase the risk of conventional cardiac surgery. The rate of delirium (acute confusional state) after surgery in these patients may exceed 50%. Estimated hospital costs associated with delirium at Toronto General Hospital last year exceeded $1-million CAD. Pain after surgery and the use of opioids (morphine type of pain-relief drugs) are known to increase the risk of delirium. The investigators plan to minimize the use of opioids and improve pain management by replacing the standard intravenous opioid-based pain management with the paravertebral nerve block using only the local anesthetic. These two management strategies will be compared with respect to the rate of delirium, duration of hospital stay, and the overall costs.

Hypothesis: Paravertebral analgesia with LA decreases the incidence of delirium after trans-apical AVR when compared to standard systemic opioid-based analgesia.

DETAILED DESCRIPTION:
A prospective, randomized, controlled, multicentre study (Toronto General Hospital and Sunnybrook Health Science Centre, Toronto, Canada.) The investigators are planning to replace the standard intravenous opioid analgesia with a continuous paravertebral block using local anesthetic after trans-apical aortic valve replacement.

Anesthesia management will be standardized to minimize any impact that anesthetic type may have on neurological outcomes.

Metrics to evaluate outcomes: Assessment of delirium will be performed utilizing the CAM-ICU preoperatively (baseline) and postoperatively every 12 hours or as needed according to the patient's condition during the first 7 postoperative days or until discharge.

The CAM recognizes both, hyperactive and hypoactive, forms of delirium. It includes four-step algorithm and assesses 1) an acute onset of changes or fluctuations in the course of mental status, 2) inattention, 3) disorganized thinking and 4) an altered level of consciousness. The patient is determined to be delirious (CAM positive) if he/she manifests both features 1 and 2, plus either feature 3 or 4.

Primary screening for delirium will be performed by the nursing staff. Diagnose of delirium will be confirmed by the psychiatry consult. Assessment of Sedation and Pain: Standardized according to institutional guidelines.

Cost Calculations: The total cost (summation of direct-variable, direct-fixed, and overhead costs) for each patient will be determined for both study groups.

ELIGIBILITY:
Inclusion Criteria:

* Consenting subjects who are scheduled to undergo the TAVI surgical procedure

Exclusion Criteria:

* patients with symptomatic cerebrovascular disease,
* history of delirium and schizophrenia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2011-06; Primary Completion 2016-06-10 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Primary Outcome: Dichotomous outcome,number of patients with delirium in the two study groups. | 2 years
  The primary objective is to determine if paravertebral analgesia with local anesthetic (LA) reduces the incidence of delirium after trans-apical AVR.

SECONDARY OUTCOMES:
Hospital length of stay | 2 years
Total cost will be compared between the two groups. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Toronto General Hospital, Toronto, Ontario, Canada